CLINICAL TRIAL: NCT06904742
Title: Clinical and Microbiological Evaluation Of The Efficacy Of Herbal Mouthwashes in Gingivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Altinbas University (Other)
Responsible Party: Principal Investigator, Candan Pelin, dentist, Altinbas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/213
Record Dates: First submitted 2025-01-27; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Periodontal Diseases
Keywords: gingivitis; essential oil; tea tree oil; thyme; qPCR
MeSH Terms: conditions — Periodontal Diseases; Gingivitis | interventions — Tea Tree Oil; Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tea Tree Oil Mouthwash Group (Active Comparator): Patients were randomized to receive the respective mouthwashes. Participants were instructed to use 15 mL of mouthwash twice-daily for one minute per application and to avoid from rinsing or consuming food for 30 minutes post-application.
  Interventions: Drug: Tea tree oil
- non-alcohol EO mouthwash group (Active Comparator): Group II; non-alcohol EO mouthwash group, patients who were administered non-alcohol essential oil mouthwash (15 mL of (Listerine Total Care Zero Mouthwash, Listerine ® for 1 min) (n=13)
  Interventions: Drug: LISTERINE ZERO Alcohol Mouthwash COOL MINT
- thyme-containing hydrosol group (Active Comparator): Group III; thyme-containing hydrosol group, of patients who were administered thyme-containing Mouthwash (15 mL of thyme hydrosol, Arifoğlu ®for 1 min) (n = 13).
  Interventions: Drug: Thyme oil hydrosol
- Control group (Placebo Comparator): placebo group, patients who were administered placebo mouthwash (15 mL of placebo mouthwash for 1 min.) (n=13)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tea tree oil — Our study's findings might have a important impact on the field of periodontology, providing valuable insights into the potential of herbal mouthwashes as an adjunct to NSPT in gingivitis treatment. A literature review reveals that regarding the mouthwash protocols, most studies mentioned use twice daily . Most studies used 10-15 ml as a dose, and rinsing time ranged from 30-90 s. In this study, similar to the literature, patients were prescribed to rinse twice daily, 15 ml for 30 s. The operator explained information about oral hygiene practices at baseline. With this approach, adequate mechanical cleaning action was obtained, and participants became more aware of importance of oral hygiene. Low scores of PI and GI in placebo group at 3rd month can be attributed to this interaction and can mask the maximum effects of herbal mouth rinses.
  Arms: Tea Tree Oil Mouthwash Group
Drug: Thyme oil hydrosol — Our study's findings might have a important impact on the field of periodontology, providing valuable insights into the potential of herbal mouthwashes as an adjunct to NSPT in gingivitis treatment. A literature review reveals that regarding the mouthwash protocols, most studies mentioned use twice daily (Santi et al., 2019). Most studies used 10-15 ml as a dose, and rinsing time ranged from 30-90 s (Santi et al., 2019). In this study, similar to the literature, patients were prescribed to rinse twice daily, 15 ml for 30 s. The operator explained information about oral hygiene practices at baseline. With this approach, adequate mechanical cleaning action was obtained, and participants became more aware of importance of oral hygiene. Low scores of PI and GI in placebo group at 3rd month can be attributed to this interaction and can mask the maximum effects of herbal mouth rinses.
  Arms: thyme-containing hydrosol group
Drug: LISTERINE ZERO Alcohol Mouthwash COOL MINT — Our study's findings might have a important impact on the field of periodontology, providing valuable insights into the potential of herbal mouthwashes as an adjunct to NSPT in gingivitis treatment. A literature review reveals that regarding the mouthwash protocols, most studies mentioned use twice daily. Most studies used 10-15 ml as a dose, and rinsing time ranged from 30-90 s . In this study, similar to the literature, patients were prescribed to rinse twice daily, 15 ml for 30 s. The operator explained information about oral hygiene practices at baseline. With this approach, adequate mechanical cleaning action was obtained, and participants became more aware of importance of oral hygiene. Low scores of PI and GI in placebo group at 3rd month can be attributed to this interaction and can mask the maximum effects of herbal mouth rinses.
  Arms: non-alcohol EO mouthwash group
Drug: Placebo — Placebo mouthwash had been used in 13 patients for 3 months
  Arms: Control group

SUMMARY:
Plaque-induced gingivitis is a clinical condition that appears to cause persistent inflammation in gingiva. It is a preliminary cause to periodontitis but it can be inverted to address the risk of periodontitis development. This randomize controlled clinical trial (RCT) aims to clinically and microbiologically evaluate the effectiveness of different herbal mouthwashes as an adjunct treatment to non-surgical periodontal therapy (NSPT) in patients with gingivitis. A total of 52 patients diagnosed with gingivitis were incorporated into the RCT and categorized into four groups as follows: Tea tree oil (Tebodont®), thyme hydrosol (Arifoglu®), essential oil (Listerine®), and placebo. The patients were advised to wash with15 ml of prescribed mouthwash twice a day for a period of 3rd months after NSPT. Clinical periodontal measurements; including plaque index (PI), gingival index (GI) and probing pocket depth (PPD) and microbiological sampling, were performed before enrollment and in 3rd months. Plaque samples were examined by quantitative polymerase chain reaction(qPCR).

DETAILED DESCRIPTION:
This randomize controlled clinical trial aims to clinically and microbiologically evaluate the effectiveness of different herbal mouthwashes as an adjunct treatment to non- surgical periodontal therapy in patients with gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* According to EFP in 2017, gingivitis patients with a PPD ≤3 mm, BOP in the whole mouth ≥ % 10 and no radiological bone loss
* Having ≥ 20 teeth
* Male or female ≥ 18 years old
* Systemically healthy patients

Exclusion Criteria:

* Using of any antioxidant or antimicrobial agent in the last 6 months

  •. Smoking
* Pregnancy
* Alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Reduction in PI | Each patient in the trial was followed up for 3rd month. During the follow up, at 30 days the patients were called to the clinic.The data were recorded at baseline and 3rd month
  PI is the amount of microbial dental plaque assesed on 6 sites of per tooth. In addition to mechanical plaque control, plaque index was our primary evaluation of the mechanism of action of mouthwashes in our study.
Reduction in GI | Each patient in the trial was followed up for 3rd month. During the follow up, at 30 days the patients were called to the clinic.The data were recorded at baseline and 3rd month
  GI introduce system for the assessment of gingival condition. For the evaluation of the index, 6 points (mesiobuccal, midpoint, distobuccal; mesiopalatinal, midpoint, distopalatinal) are examined according to the presence of bleeding that occurs after the examination with the probe and index values between 0-3 are given.
Reduction in Bleeding on Probing | Each patient in the trial was followed up for 3rd month. During the follow up, at 30 days the patients were called to the clinic.The data were recorded at baseline and 3rd month
  Bleeding on probing is one of the important parameters in the diagnosis of gingivitis, reduction in bleeding on probing is the primary outcomed.

SECONDARY OUTCOMES:
Reduction in PPD | Each patient in the trial was followed up for 3rd month. During the follow up, at 30 days the patients were called to the clinic.The data were recorded at baseline and 3rd month
  PPD is an important parameter in the evaluation of the treatment of periodontal diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Altinbas University, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided